CLINICAL TRIAL: NCT01039233
Title: Randomized, Bioequivalence Study of Bicalutamide 50 mg Tablet and Casodex 50 mg Tablet Following a 50 mg Dose in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Bicalutamide 50 mg Tablet and Casodex 50 mg Tablet in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kremers Urban Development Company (Industry)
Collaborators: Watson Laboratories, Inc. (Industry)
Responsible Party: Richard Larouche, M.D., Medical Director, sfbc Anapharm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50013
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Bioequivalency
MeSH Terms: interventions — bicalutamide; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bicalutamide 50 mg Tablet (Experimental)
  Interventions: Drug: Bicalutamide 50 mg Tablet vs Casodex® 50 mg Tablet
- Casodex® 50 mg Tablet (Active Comparator)
  Interventions: Drug: Bicalutamide 50 mg Tablet vs Casodex® 50 mg Tablet

INTERVENTIONS:
Drug: Bicalutamide 50 mg Tablet vs Casodex® 50 mg Tablet

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of bicalutamide 50 mg tablet (test) versus Casodex (reference), administered as 1 x 50 mg tablet under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Male, non-smoker, 18 years of age and older;
* Capable of consent;
* BMI≥19.0 and <30.0 kg/m2.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins. garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 6 months preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:

  * 50 mL to 300 mL of whole blood within 30 days,
  * 301 mL to 500 mL of whole blood within 45 days, or
  * more than 500 mL of whole blood within 56 days prior to drug administration.

Ages: 20 Years to 73 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-05; Primary Completion 2005-06 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration) | 144 hour
AUC0-inf area under the concentration-time curve from time zero to infinity) | 144 hour
Cmax (maximum observed concentration of drug substance in plasma) | 144 hour

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D., Principal Investigator — SFBC Anapharm
Locations (1):
- SFBC Anapharm, Montreal, Quebec, Canada